CLINICAL TRIAL: NCT00197093
Title: A Placebo Controlled, Double-Blind, Randomised Study Investigating the Safety, Tolerability and Pharmacokinetics of Ascending Multiple Oral Doses of SB-773812 in Male and Female Schizophrenic Patients for up to 28 Days
Brief Title: In-Patient Study In Schizophrenic Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 773812/003
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2009-05-18 (Estimated); Status verified 2009-05

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; safety; tolerability; pharmacokinetics
MeSH Terms: conditions — Schizophrenia

INTERVENTIONS:
Drug: SB773812

SUMMARY:
This study is a placebo-controlled study to assess the safety and tolerability of a novel antipsychotic medication, (773812) when given to schizophrenic patients for twenty-eight days. Assessments include blood sampling to determine drug concentrations, psychiatric assessments while under treatment, and movement assessments to evaluate potential side effects.

ELIGIBILITY:
Inclusion Criteria:

* Must have schizophrenia that has been stable for at least three months.
* Willing to discontinue current anti-psychotic medications (under supervision) prior to the study.
* Willing to live at the study center for a total of 38 days and then return for three follow-up visits.

Exclusion Criteria:

* Taking medications for conditions other than schizophrenia.
* History of alcohol or drug abuse within six months of the study, and their alcohol consumption must meet moderate guidelines.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60
Dates: Start 2004-09

PRIMARY OUTCOMES:
Safety and Tolerability of 773812 during 28 days of dosing. Pharmacokinetics of 773812 after repeat dosing.

SECONDARY OUTCOMES:
Assessment of (1) changes in testing scores on a range of psychiatric assessments (PANSS, BPRS. CGI) (2) psychometric performance and (3)body weight/ girth measurement /glucose and lipd measurement, each as a function of duration of dosing.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline